CLINICAL TRIAL: NCT04179383
Title: Identification of Reversible Cerebral Vasoconstriction Syndrome's Precipitating Factors. Triggers And Risk Factors to Develop a Reversible Cerebral Vasoconstriction Syndrome
Brief Title: Triggers And Risk Factors to Develop a Reversible Cerebral Vasoconstriction Syndrome
Acronym: TARDIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9894
Record Dates: First submitted 2018-11-29; First posted 2019-11-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Reversible Cerebral Vasoconstriction Syndrome
Keywords: Thunderclap headache
MeSH Terms: conditions — Headache Disorders, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Other): Patient presenting a Reversible Cerebral Vasoconstriction Syndrome (RCVS) :
  * Questionnaires about anxiety, depression ;
  * Constitution of a biobank (if specific consent) at inclusion and at 3 months
  Interventions: Other: Constitution of a biobank
- Volunteers (Other): Volunteers admitted for a non neurological or non vascular pathology or healthy volunteers accompanying a patient :
  * Questionnaires about anxiety, depression ;
  * Constitution of a blood biobank (if specific consent)
  Interventions: Other: Constitution of a biobank

INTERVENTIONS:
Other: Constitution of a biobank — We are collecting additional blood and CSF samples for patients (during RCVS episode and after resolution of RCVS episode) and for control subjects to constitute a biobank, in order to compare different biologic parameters between RCVS patients and healthy volunteers. A specific agreement will be asked to patients and control subjects before collection of samples.
  This is why this study is classified as 'interventional' rather than 'observational'.

SUMMARY:
This study will be the first to evaluate the role played by potential precipitating factors and risk factors in Reversible Cerebral Vasoconstriction Syndrome (RCVS) through of prospective selection of carefully characterised patients and controls. The impact of these factors on the prognosis will be evaluated through a follow-up assessment of patients.

Our study will include the formation of a clinicoradiological database and a biobank (plasma, cerebro-spinal fluid, DNA) which will be the tools of a future large multicentre study on RCVS.

DETAILED DESCRIPTION:
Introduction : Reversible Cerebral Vasoconstriction Syndrome (RCVS) combines headaches and segmental constriction of cerebral arteries that resolves within 3 months.

It is the most recurrent reason of cerebral arteriopathy in people under 70 and of thunderclap headache in absence of aneurysmal subarachnoid haemorrhage.

Objectives :

* Principal: identify RCVS's precipitating factors
* Secondary:

  1. Determine if migraine, anxiety, depression are risk factors of RCVS.
  2. Determine the role of precipitating factors and risk factors on the RCVS's prognosis in short, medium and long term.
  3. Start a formation of a large clinicoradiological database and a biobank (plasma, cerebro-spinal fluid, DNA).

Methodology :

Monocentric analytic observational 'Case - Control' study with prospective inclusion of cases in a follow-up cohort.

This type of study is nevertheless considered interventional because we are collecting additional blood and CSF samples to constitute a biobank.

ELIGIBILITY:
Inclusion criteria:

* For the Patients

  * Men and women of 18 and more years old
  * Taken care in the CHU of Montpellier
  * Diagnosis of SVCR or SVCR without visible vasoconstriction makes in 14 days preceding the inclusion
  * According to the consensual criteria of diagnosis and those of the international classification of the headaches ICHD-3
  * Informed consent and writes for the participation in the study
* For volunteers

  * Men and women of 18 and more, mated in the Cases on the sex and the age
  * Patients with an acute pathology not Neurological and not vascular (for example, eye foreign body) OR Healthy Subjects
  * Informed written consent and for the participation in the study

Exclusion criteria:

* Coma, insanity, language barrier or severe aphasia preventing from answering the questions
* Follow-up considered impossible for 3 months (e.g.: priority associated pathology in the care, the transfer(transformation))
* People placed under legal protection
* Refusal to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Presence of, at least, one assumed trigger or risk factors | 3 months
  The relationship between the assumed precipitating factors and RCVS will be evaluated by comparing the frequencies of exposure of suspected precipitating factors between cases and controls, and given by calculating an odds ratio.
  The assumed trigger or risk factors are : a physical and / or emotional stress within 30 days before the clinical beginning; presence of chronic neurological or psychiatric disease (migraine, primary thunderclap headache or circumstancial headache, anxiety or depression); vascular risk factors; and hormonal status in women.

SECONDARY OUTCOMES:
Comparison between precipitating factors and clinico-radiological manifestations of RCVS | 3 months
  Evaluation of Clinical manifestations (headache, seizures, focal neurological deficit) according to the presence of precipitating factors
Comparison between precipitating factors and clinico-radiological manifestations of RCVS | 3 months
  Evaluation of Brain lesion (stroke, posterior reversible encephalopathy syndrome) according to the presence of precipitating factors
Comparison between precipitating factors and clinico-radiological manifestations of RCVS | 3 months
  Evaluation of Severity of cerebral arteries' vasoconstriction, according to the presence of precipitating factor
Comparison between precipitating factors and clinico-radiological manifestations of RCVS | 3 months
  Evaluation of Lesion of intracranial and / or cervical arteries, according to the presence of precipitating factors
Comparison between precipitating factors and clinico-radiological manifestations of RCVS | 3 months
  Evaluation of Modified Rankin Score, evaluated 3 month after clinical beginning, according to the presence of precipitating factors.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas CORTI, Principal Investigator — CHU de Montpellier
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No